CLINICAL TRIAL: NCT04705623
Title: A Single-center, Randomized, Controlled, Open-labelled, Two-armed, Interventional Clinical Trial Investigating the Effect of a 12 Week Iyengar Yoga Intervention on the Bio-functional Age of Postmenopausal Women.
Brief Title: Influence of Iyengar Yoga on the Bio-functional Age of Postmenopausal Women
Acronym: IIYBFAPW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-01794
Record Dates: First submitted 2020-12-30; First posted 2021-01-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Postmenopausal; Postmenopausal Flushing
Keywords: Biofunctional age; Yoga

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, controlled, open-labelled, two-armed, interventional clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group receives weekly 90 minute yoga classes over a course of 12 weeks. They are also asked to do two 45-minute yoga classes at home each week and document these in a Diary.
  Interventions: Behavioral: Iyengar Yoga
- Control (No Intervention): The control group receives an assessment of their biofunctional status at the beginning and the end of the study (same as the intervention group).

INTERVENTIONS:
Behavioral: Iyengar Yoga — Weekly 90 minute Iyengar Yoga classes taught y a professional instructor. Twice weekly 45 minute self practice of Iyengar Yoga at home by the participants
  Arms: Intervention

SUMMARY:
The purpose of this Study is to find out if Iyengar-Yoga has a rejuvenating effect on women after menopause. The biofunctional status of the study participants will be assessed before and after a 12-week yoga program.

DETAILED DESCRIPTION:
Postmenopausal women qualifying as participants for the study are patients at the Universitätsklinik für Frauenheilkunde in Bern or are recruited through public advertisement. After giving informed consent the patients will be screened for inclusion and exclusion criteria and their biofunctional Status will be assessed. The participants of the study will then be randomly assigned to the intervention group (12 week yoga program) or to the control group. In addition to the 90 minutes yoga sessions instructed by a professional yoga teacher, the participants of the intervention group are asked to perform two yoga sessions lasting 45 minutes per week at home and document these in a diary.

After the 12 weeks the biofunctional Status of all participants of the study will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Women after Menopause (defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40mlU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy)
* Age over 18 years
* At least 4 hot flushes per day (examined through the Menopause rating scale MRS-II)
* No regular yoga practice for two years
* German as native language
* Willing to participate in 12 yoga classes as well as two 45 self practice sessions per week
* Willing to assess biofunctional Status and give blood samples

Exclusion Criteria:

* Acute and/or serious disease in the past two years (e.g. Cancer, major surgery)
* Autoimmune or chronic inflammatory disease (e.g. rheumatism, thyroid dysfunction)
* Mental illness (e.g. Depression or anxiety disorder (HADS >8))
* Acute or chronic back pain or herniated vertebral disc
* Compulsion to participate in the trial
* Attendance of less than 10 yoga lessons out of 12.
* Hormone replacement therapy (HRT)
* Smoking > 20 Cigarettes per day or over 20 packyears
* Consumption of >30g alcohol per day (>1 liter of beer or >0.3 dl of wine)
* Previous periodic participation in yoga classes within the last two years
* Inability or contraindications to undergo the investigated intervention
* Participants incapable of judgement or participants under tutelage Diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participation is only possible for biologically female human beings
Enrollment: 72 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Decrease of the biofunctional age (BFA) through a 12 week Iyengar yoga intervention compared to the control group with no yoga classes. In order to evaluate the BFA a biofunctional Status (BFS) has to be assessed. | 12 weeks
  The BFS is a generic, age- and sex-specific test battery comprising holistic characteristics from physical, mental-emotional and social areas. The single values of the BFS test battery were scaled and differentiated for chronological age (CA) and sex. Their summation makes up the so-called Bio-functional Age Index BFAI (BFAI = Σ (B-X/B-L)n/n). The BFAI is a relative measure compared to a reference population, out of which norm charts were developed. By definition, the reference population's BFAI is identical with its CA. A BFAI of an individual may be transformed into BFA (years) by means of gerontologic aging tables. This BFA (years) relates to the mean value of a certain CA. The BFA is based on a sex-specific regression and factor analysis of functional age (Mathieu et al., 2018. Illness perception in overweight and obesity and impact on bio-functional age. Archives of gynecology and obstetrics, 298(2), p. 417)

SECONDARY OUTCOMES:
Hot flushes | 12 weeks
  Change of the climacteric symptom hot flushes (number per day) measured at the beginning and after 12 weeks of the intervention
Level of High sensitive C-reactive protein (HS-CRP) | 12 weeks
  Change of the climacteric symptom Level of HS-CRP (mg/l) measured at the beginning and after 12 weeks of the intervention
Oxidative balance | 12 weeks
  Change of the climacteric symptom oxidative balance measured at the beginning and after 12 weeks of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, Prof. Dr. med, Principal Investigator — Universitätsklinik für Frauenheilkunde Bern
Locations (1):
- Dep. of Obstetrics and Gynecology, Bern University Hospital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Public access to the full protocol, patient dataset and statistical code will not be granted. The principal investigator will have ultimate authority over all of the activities.